CLINICAL TRIAL: NCT00031486
Title: A Phase III Double-Blind, Placebo-Controlled Trial of Long Term Therapy of Herpes Simplex Encephalitis (HSE): An Evaluation of Valacyclovir (CASG-204)
Brief Title: Long Term Treatment of Herpes Simplex Encephalitis (HSE) With Valacyclovir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98-022; CASG 204; N01AI30025C; N01AI30025 (NIH); NCT00001124 (obsolete NCT alias)
Record Dates: First submitted 2002-03-06; First posted 2002-03-07 (Estimated); Results first posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2011-10

CONDITIONS: Encephalitis
Keywords: encephalitis, herpes simplex, valacyclovir
MeSH Terms: conditions — Encephalitis; Herpes Simplex | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Valacyclovir (Experimental)
  Interventions: Drug: Valacyclovir
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — Valacyclovir is a L-valyl ester of acyclovir. Valacyclovir is provided in 500 mg tablets, 4 tablets (500 mg tablets) 3 times a day (every 8 hours) for 90 days.
  Arms: Valacyclovir
Drug: Placebo — Placebo (identical to active drug in appearance) 500 mg tablets, 4 tablets 3 times daily for 90 days.
  Arms: Placebo

SUMMARY:
This study involves patients 12 years and older who have been diagnosed with herpes simplex encephalitis (HSE) by a specific laboratory test and have completed treatment or are being treated with intravenous (given through a needle inserted into a vein) acyclovir. The purpose of the study is to determine if treatment with 4 tablets, 500 milligrams each, of valacyclovir given 3 times daily by mouth for 90 days is both effective and safe after completing intravenous acyclovir treatment and if it can increase survival with or without mild impairment of the brain and mental functions. Participants will be assigned to either drug or placebo (inactive substance) randomly (by chance). Study procedures will include blood samples and lumbar punctures (procedure in which a needle is inserted into the lower back to collect cerebral spinal fluid). Subjects will participate for up to 24 months.

DETAILED DESCRIPTION:
Herpes simplex encephalitis (HSE) remains the most common cause of sporadic fatal encephalitis in the world. This study is a phase III, double-blind, placebo controlled study of long term therapy with valacyclovir as a treatment of herpes encephalitis. The primary objective of this study is to assess the impact of valacyclovir (VACV) therapy (following standard intravenous acyclovir therapy) on neuropsychological impairment at one year post therapy, based on the cumulative scores of the Mattis Dementia Rating Scale (MDRS). The secondary objectives of the study are to: assess the effect of therapy on neuropsychological impairment at various time points; assess the effect of therapy on quality of life, based on the SF-36 Quality of Life Assessment; measure the effect of therapy on herpes simplex virus (HSV) deoxyribonucleic acid (DNA) in the cerebral spinal fluid (CSF); and assess the safety and tolerability of long term VACV therapy in patients with HSE. The tertiary objective of the study is to determine the frequency of symptomatic relapse/recurrence of HSE. Study participants will include 120 males and females, 12 years of age and older, diagnosed with HSE; laboratory confirmed CSF positive for HSV DNA by polymerase chain reaction (PCR). Consenting study participants will be randomized (1:1) to either valacyclovir (active drug), 500 mg tablets, four tablets three times daily for 90 days or placebo (identical to active drug in appearance), 500 mg tablets, four tablets three times daily for 90 days. The primary endpoints of the study are to assess the impact of valacyclovir therapy [following standard intravenous acyclovir (ACV) therapy] on neuropsychological impairment at one year post therapy and survival with no or mild neuropsychological impairment at 12 months after initiation of study medication, as measured by the MDRS. The secondary endpoints include: survival with no or mild neuropsychological impairment at 90 days and at 6, 12 and 24 months, as measured by the MDRS, the Mini-Mental Status Examination (MMSE), and the Glasgow Coma Scale; effect of study medication on quality of life measurements; effect of antiviral therapy on HSV DNA in CSF (measured quantitatively by PCR at Day 0 and Day 90); and safety and tolerance of VACV administered at a dose of 2.0 grams given orally three times a day for 90 days. Each study participant will participate for approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and/or assent must be obtained from the patient or legal guardian.
* Patients with encephalopathy consistent with herpes simplex encephalitis (HSE) whose cerebral spinal fluid (or brain biopsy sample) is positive for herpes simplex virus (HSV) deoxyribonucleic acid (DNA) by polymerase chain reaction (PCR).
* Patients who are receiving and will have completed intravenous (IV) acyclovir (ACV) therapy for a minimum duration of 14 days to a maximum of 21 days and a minimum dose of 30 mg/kg/day to a maximum of 60 mg/kg/day, or equivalent dose as adjusted for renal dysfunction.
* Patient is expected to be available for follow-up visits of study drug administration and through the 24 month study visit.
* Patients who are 12 years of age or older.
* Patients who weigh greater than or equal to 45.5kg (100 pounds).
* All female patients with childbearing potential must have a negative pregnancy test within 72 hours prior to initiation of study drug. If the pregnancy test is positive, the patient is ineligible for the study.
* Women must be post-menopausal, surgically sterile or willing to use adequate contraception (barrier method with spermicide, intrauterine device (IUD), oral contraceptives, implant or other licensed hormone method) from time of study enrollment through 1 month after the last dose of study treatment.
* Men must be surgically sterile or willing to use contraception (barrier method with spermicide) from time of study enrollment through 1 month after the last dose of study treatment.

Exclusion Criteria:

* Patients with herpes simplex virus (HSV) meningitis only, without evidence of HSV encephalitis.
* Patients with an anticipated life expectancy < 90 days.
* Patients with creatinine clearance of less than or equal to 50ml/min./1.73 m^2.
* Pregnant or breastfeeding females.
* Patients who have received any anti-herpesvirus medication (e.g. ganciclovir) other than intravenous acyclovir (ACV) for acute therapy of the current episode of herpes simplex encephalitis (HSE).
* Patients who are unable to swallow oral medications at the time of study drug randomization (Day 0).
* Patients who are > 3 days beyond completion of treatment course with intravenous (IV) ACV.
* Patients who are expected to receive long-term (> 30 days/year) therapy with antiviral medications active against HSV [e.g. ACV, valacyclovir (VACV), famciclovir].

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2000-09; Primary Completion 2010-06 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center - Barrow Neurological Institute - Phoenix, Phoenix, Arizona
  - University of California Davis Medical Center, Sacramento, California
  - University of Colorado, Denver, Colorado
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University Hospital - School of Medicine - Department of Neurology & Psychiatry, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Toledo, Toledo, Ohio
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (2):
  - University of Manitoba - Medical Microbiology and Infectious Diseases, Winnipeg, Manitoba
  - Kingston General Hospital - Internal Medicine - Neurology, Kingston, Ontario
- Sweden (5):
  - University of Gothenburg - Sahlgrenska Academy, Gothenberg
  - niversity of Lund - Infectious Disease, Lund
  - Karolinska University Hospital, Huddinge, Stockholm
  - Umea University - Infectious Diseases, Umeå
  - Uppsala University Hospital, Uppsala
- University College London - Royal Free Campus - Virology, London, United Kingdom

REFERENCES:
- [Derived] Gnann JW Jr, Skoldenberg B, Hart J, Aurelius E, Schliamser S, Studahl M, Eriksson BM, Hanley D, Aoki F, Jackson AC, Griffiths P, Miedzinski L, Hanfelt-Goade D, Hinthorn D, Ahlm C, Aksamit A, Cruz-Flores S, Dale I, Cloud G, Jester P, Whitley RJ; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Herpes Simplex Encephalitis: Lack of Clinical Benefit of Long-term Valacyclovir Therapy. Clin Infect Dis. 2015 Sep 1;61(5):683-91. doi: 10.1093/cid/civ369. Epub 2015 May 8. PMID 25956891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled in the study presented with findings of HSE.
Pre-assignment Details: Patients considered for enrollment are those who are receiving and will have completed IV Acyclovir for a minimum duration of 14 days to a maximum of 21 days at a minimum dose of 30 mg/kg/day to a maximum dose of 60 mg/kg/day.
Groups:
- Valacyclovir: four 500 mg tablets 3 times a day for 90 days
- Placebo: four placebo tablets (identical to active drug in appearance) 3 times a day for 90 days
Period: Overall Study
Arm/Group | Valacyclovir | Placebo
Started | 40 | 47
Completed | 33 | 35
Not Completed | 7 | 12
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Death | 0 | 3
Not completed — Non-compliant | 0 | 4
Not completed — Did not meet eligibility requirement | 2 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 40 | 47 | 87
Age Continuous [Mean (Inter-Quartile Range); unit: years] | 53.5 [14 to 77] | 56 [26 to 83] | 55 [14 to 83]
Age, Customized [Number; unit: participants]
  12-18 years | 2 | 0 | 2
  19-40 years | 7 | 5 | 12
  41-60 years | 18 | 22 | 40
  61 years or older | 13 | 20 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 20 | 27 | 47
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17
  Canada | 6 | 4 | 10
  United Kingdom | 0 | 3 | 3
  Sweden | 26 | 31 | 57

OUTCOME MEASURES:

1. Primary Outcome: Survival With no or Mild Neuropsychological Impairment at 12 Months After Initiation of Study Medication as Measured by the Mattis Dementia Rating Scale (MDRS)
Description: Number of subjects who were assessed to have no or mild neuropsychological impairment at 12 months using the Mattis Dementia Rating Scale. (A score of 121 or higher refects no or mild neuropsychological impairment.) Scale is: 139-144 normal; 121-139 mild; 114-120 moderate; 87-113 severe; and <=86 very severe.
Time Frame: One year post therapy.
Population: All subjects that survived to 12 months and were assessed.
Measure: Number; unit: Participants
Groups:
- Valacyclovir: four 500 mg tablets taken 3 times a day for 90 days
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 33 | 36 | 62
Participants
  MDRS Score >= 121 (positive) | 28 | 34 | 62
  MDRS score < 121 (negative) | 5 | 2 | 7

2. Secondary Outcome: Effect of Study Medication on Quality of Life Measurements.
Description: The SF-36 Questionnaire measures quality of life as reported by the subject. The questionnaire contains 36 questions, each questions can be assigned a maximum score of 100. For each subject, a perfect score would be 3600, hence the higher score is best. The calculated scores reported in the table below reflect the diffence between Day 0 (day study drug started) and Day 90, Day 0 (day study drug started) and Month 6, and Day 0 (day study drug started) and Month 12.
Time Frame: Day 0 and 90, Day 0 and Month 6 and Day 0 and Month 12
Population: All subjects that were assessed at baseline and the following time points: 90 days, 6 and 12 months.
Measure: Median (Full Range); unit: Scores on a scale Change in SF-36
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 28 | 33 | 61
Scores on a scale Change in SF-36
  SF-36 score difference from day 0 to 90 | 465 [-745 to 2360] | 307.5 [-935 to 2575] | 355 [-935 to 2575]
  SF-36 score difference from day 0 to 6 months | 722.5 [-1060 to 2125] | 475 [-1170 to 2215] | 635 [-1170 to 2215]
  SF-36 score difference from day 0 to 12 months | 1095 [-1565 to 2240] | 985 [-1330 to 2355] | 985 [-1565 to 2355]

3. Secondary Outcome: Effect of Antiviral Therapy on Herpes Simplex Virus (HSV) Deoxyribonucleic Acid (DNA) in Cerebral Spinal Fluid (CSF)
Description: Few CSF specimens were collected on day 90, hence unable to calculate the difference in PCR at day 0 and day 90.[measured quantitatively by polymerase chain reaction (PCR)].
Time Frame: Day 0 and Day 90.
Population: The number of participants analyzed is 0 because there specimens obtained were inadequate and insufficient to analyze.
Measure: Number; unit: viral load
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Median Number of Reported AEs Describing Safety and Tolerance of Valacyclovir (VACV), Evaluated by the Number Adverse Events, Administered at a Dose of 2.0 Grams Given Orally 3 Times a Day for 90 Days.
Description: The measure is the number of adverse events per subject. Adverse events were recorded from time of first dose of study drug through 6 months post start of study drug.
Time Frame: 6 months
Measure: Median (Full Range); unit: Events per participants
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 36 | 42 | 78
Events per participants | 8.5 [1 to 25] | 8 [1 to 38] | 8 [1 to 38]

5. Secondary Outcome: Survival With no or Mild Neuropsychological Impairment at 90 Days and at 6 and 12 Months, as Measured by the Mattis Dementia Rating Scale (MDRS)
Description: The assessment scoring for the Mattis Dementia Rating Scale is as follows: 139 - 144: no neuropsychological impairment; 121- 138: mild neuropsychological impairment; 114 - 120: moderate neuropsychological impairment; 87 - 113: severe neuropsychological impairment; and <=86: very severe neuropsychological impairment.
Time Frame: 90 days, 6 and 12 months
Population: All subjects that survived and were assessed at 90 days, 6 and 12 months.
Measure: Number; unit: Participants
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 31 | 36 | 67
Participants
  MDRS score >= 121 (90 days) | 28 | 31 | 59
  MDRS score < 121 (90 days) | 3 | 5 | 8
  MDRS score >= 121 ( 6 months) | 24 | 31 | 55
  MDRS score < 121 (6 months) | 5 | 4 | 9
  MDRS score >= 121 (12 months) | 28 | 34 | 62
  MDRS score < 121 (12 months) | 5 | 2 | 7

6. Secondary Outcome: Survival With no or Mild Neuropsychological Impairment at 90 Days, and at 6 and 12 Months, as Measured by the Mini-Mental Status Examination (MMSE).
Description: The assessment score for the Mini-Mental Status Examination is as follows: 27 - 30: no neuropsychological impairment; 23 - 26: mild neuropsychological impairment; 16 - 22: moderate neuropsychological impairment; 11 - 15 severe neuropsychological impairment; and <=10: very severe neuropsychological impairment.
Time Frame: 90 days, 6 and 12 months
Population: All subjects that survived and were assessed at 90 days, 6 and 12 months.
Measure: Number; unit: Participants
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 29 | 36 | 65
Participants
  MMSE score >= 23 (90 days) | 26 | 31 | 57
  MMSE score < 23 (90 days) | 3 | 5 | 8
  MMSE score >= 23 (6 months) | 23 | 29 | 52
  MMSE score < 23 (6 months) | 4 | 4 | 8
  MMSE score >= 23 (12 months) | 28 | 30 | 58
  MMSE score < 23 (12 months) | 4 | 5 | 9

7. Secondary Outcome: Survival With no or Mild Neuropsychological Impairment at 90 Days and at 6 and 12 Months, as Measured by the Glasgow Coma Scale (GCS).
Description: The assessment scoring for the Glasgow Coma Scale is as follows: 15: no neuropsychological impairment; 12 - 14: mild neuropsychological impairment; 9 - 11: moderate neuropsychological impairment; 6 to 8: severe neuropsychological impairment; and <6: very severe neuropsychological impairment.
Time Frame: 90 days, 6 and 12 months
Population: All subjects that survived and were assessed at 90 days, 6 and 12 months.
Measure: Number; unit: Participants
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 33 | 37 | 70
Participants
  GCS score >= 12 (90 days) | 30 | 37 | 67
  GCS score < 12 (90 days) | 0 | 0 | 0
  GCS score >= 12 (6 months) | 31 | 36 | 67
  GCS score < 12 (6 months) | 0 | 0 | 0
  GCS score >= 12 (12 months) | 33 | 37 | 70
  GCS score < 12 (12 months) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Valacyclovir | Placebo
Serious Adverse Events (participants affected / at risk) | 16/40 | 29/47
Other Adverse Events (participants affected / at risk) | 36/40 | 39/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=40) | Placebo (N=47)
Agitated depression (Psychiatric disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Billiary dyskinesia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 2 (3) | 3 (4)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Encephalitis (Nervous system disorders) | 1 (1) | 1 (1)
Encephalitis herpes (Infections and infestations) | 1 (1) | 2 (2)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lymphadenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Retinal ischaemia (Eye disorders) | 1 (1) | 0 (0)
Simple partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valacyclovir (N=40) | Placebo (N=47)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ageusia (Nervous system disorders) | 2 (2) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (2)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0)
Alanine aminotransferase abnormal (Investigations) | 1 (1) | 1 (2)
Alanine aminotransferase decreased (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Amnesia (Nervous system disorders) | 1 (2) | 0 (0)
Anosmia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (5) | 3 (4)
Aphasia (Nervous system disorders) | 0 (0) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0)
Blood creatinine abnormal (Investigations) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 3 (4) | 2 (3)
Blood glucose abnormal (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 2 (2)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Blood urea (Investigations) | 1 (1) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1)
Blood uric acid abnormal (Investigations) | 1 (1) | 0 (0)
Blood uric acid decreased (Investigations) | 1 (1) | 1 (1)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 1 (2) | 0 (0)
Candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (3)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Convulsion (Nervous system disorders) | 1 (1) | 6 (9)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 7 (8) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (4)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (5) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dyscalculia (Nervous system disorders) | 0 (0) | 1 (1)
Dysesthesia extremity (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (2)
Encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Encephalitis herpes (Infections and infestations) | 2 (2) | 1 (1)
Eosinophil count abnormal (Investigations) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (2)
Extensor plantar response (Nervous system disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 6 (6) | 6 (7)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Genital candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Genital infection (Infections and infestations) | 0 (0) | 1 (1)
Gingival hyperplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Global anmesia (Nervous system disorders) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 2 (3)
Haematocrit abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hallucinaion (Psychiatric disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 12 (14) | 7 (10)
Hepatic enzyme increased (Investigations) | 0 (0) | 3 (3)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hyperreflexia (Nervous system disorders) | 2 (2) | 0 (0)
Hypertonia (Nervous system disorders) | 1 (2) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 1 (1)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Injection site vesicles (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 6 (6)
Irritability (General disorders) | 2 (2) | 1 (1)
Leg paresis (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Mental status change (Psychiatric disorders) | 0 (0) | 1 (2)
Meralgia paraesthetica (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (20) | 12 (18)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Neutrophil count abnormal (Investigations) | 1 (1) | 0 (0)
Nightmares (Psychiatric disorders) | 1 (1) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1) | 1 (1)
Obsessive-compulsive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (3)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Protein urine present (Investigations) | 0 (0) | 1 (1)
Pyloric abscess (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 5 (5)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Red blood cell count abnormal (Investigations) | 1 (1) | 0 (0)
Reticulocyte count abnormal (Investigations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 1 (1) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (3) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 3 (3) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (3)
Urinary tract infection (Infections and infestations) | 7 (11) | 5 (6)
Urine analysis abnormal (Investigations) | 1 (2) | 0 (0)
Urine leukocyte esterase (Investigations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 3 (4)
Weight increased (Investigations) | 1 (1) | 0 (0)
White blood cells urine positive (Investigations) | 2 (3) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No